CLINICAL TRIAL: NCT04813302
Title: Influence of Anatomical Factors Upon Root Coverage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Gonzalo Blasi, Clinical Instructor, Universitat Internacional de Catalunya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PER-ECL-2019-04
Record Dates: First submitted 2021-03-21; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Gingival Recession; Gingival Diseases; Periodontal Attachment Loss
MeSH Terms: conditions — Gingival Recession; Gingival Diseases; Periodontal Attachment Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gingival recession treatment (Experimental): Gingival recession treatment by means of a coronally advanced flap and a connective tissue graft
  Interventions: Procedure: Coronally advanced flap and connective tissue graft

INTERVENTIONS:
Procedure: Coronally advanced flap and connective tissue graft — CAF+CTG treatment will be performed by starting with two vertical releasing incisions lateral to the teeth to be treated and split-full-split thickness flap will be raised beyond the MGJ. The periosteum will be cut, and a blunt dissection into the vestibular lining mucosa will be carried out to eliminate muscle tension so that the mucosal flap can be passively positioned above the level of CEJ on the tooth. The papillae adjacent to the involved teeth will be de-epithelialized. CTG of 1mm in thickness will be harvested from the posterior palate by means of disepithelization of a free gingival graft, cut to the exact size of the defect, and placed over the dehisced defect, sutured to the interdental papillae and subsequently covered with CAF. Sling sutures will be placed to stabilize the flap in a coronal position about 1-2 mm above the CEJ , followed by interrupted sutures to close the releasing incisions.

SUMMARY:
Introduction:

Gingival recession is a lesion characterized by the loss of attachment of root surface of the tooth, resulting in an apical migration of the gingival margin that occasionally generates aesthetic problems, hypersensitivity and difficulty in maintaining proper hygiene.

Several anatomical factors have been associated both with the incidence and progression of gingival recession and with the prognosis of the surgical treatments proposed for its correction. These factors include the absence of keratinized tissue, the gingival phenotype, root prominence and shallow vesrtibular depth.

Objectives:

The objective of the study is to evaluate, through a series of prospective cases, the influence of each of the anatomical factors on the success of root coverage.

Methods:

20 patients with gingival recession defects will be treated with CAF+CTG using various autogenous gingival graft. Three-dimensional analysis of superimposed preoperative and postoperative images will be performed. Linear and surface root coverage will be calculated and correlated to various anatomical parameters such as vestibular depth and root prominence. A multilevel statistical analysis will be conducted, adjusting for the correlation among multiple observations.

DETAILED DESCRIPTION:
- Pre-surgical treatment: Initial periodontal therapy will be performed 1 month prior to surgery. Patients will receive a pre-surgical prophylaxis, oral hygiene instructions and elimination of toothbrushing traumatic technique, if needed. They will be taught to use a toothbrush of medium hardness applying Roll brushing technique.

- Surgical treatment: In brief description, CAF+CTG treatment will be performed by starting with two vertical releasing incisions lateral to the teeth to be treated and split-full-split thickness flap will be raised beyond the MGJ. The periosteum will be cut, and a blunt dissection into the vestibular lining mucosa will be carried out to eliminate muscle tension so that the mucosal flap can be passively positioned above the level of CEJ on the tooth. The papillae adjacent to the involved teeth will be de-epithelialized and the exposed root surfaces will be treated with pre-conditioning EDTA (Straumann PrefGel®) for 2 minutes. CTG of 1mm in thickness will be harvested from the posterior palate by means of disepithelization of a free gingival graft (22), cut to the exact size of the defect, and placed over the dehisced defect, sutured to the interdental papillae (7-0 Polyglactin 910, Vycril, Ethicon, Johnson and Johnson, New Brunswick, NJ, USA) and subsequently covered with CAF. Sling sutures will be placed to stabilize the flap in a coronal position about 1-2 mm above the CEJ (6-0 Polypropylene, Prolene, Ethicon, Johnson and Johnson, New Brunswick, NJ, USA), followed by interrupted sutures to close the releasing incisions.

Patients will be instructed to avoid any mechanical trauma or tooth brushing in the surgical sites for 2 weeks. Analgesic medication (ibuprofen) will be prescribed as required and patients will be instructed to rinse with Chlorhexidine three times per day for 2 weeks. Sutures will be removed after 14 days. Two weeks after surgery, patients will resume mechanical tooth cleaning with a soft toothbrush. Patients will be recalled at 1, 3 and 6 months for professional oral hygiene procedures.

- Post-surgical instructions and infection control: Patients will be instructed to avoid any mechanical trauma or tooth brushing in the surgical sites for 2 weeks. Analgesic medication (ibuprofen) will be prescribed as required and patients will be instructed to rinse with Chlorhexidine 0.12% two times per day for 2 weeks. Sutures will be removed after 14 days. Two weeks after surgery, patients will resume mechanical tooth cleaning with a soft toothbrush. Patients will be recalled at 1, 3 and 6 months for professional oral hygiene procedures.

- Data collection: A guidebook will be prepared to systematize the procedures for sample and data collection. The data will be later transferred to a computerized database (Epidata®, Odense, Denmark, Europe).

A) Sociodemographic data An interview will be conducted during the pre-surgical visit to obtain information regar- ding age, sex, medical history, use of medication, exposure to tobacco, pregnancy and previous periodontal surgeries.

B) Clinical measurements Probing depth (PD) and keratinized tissue width (KTW) will be measured using a periodontal probe (PCP UNC 15, Hu-Friedy, Chicago, IL, USA). KTW will be measured at the most apical point in the GM to the mucogingival junction at the mid-buccal site to the nearest millimeter. KTT will be measured 1.5mm and 3mm apical to the GM using an injection needle, perpendicular to the tissues surface and a silicon stop over the gingival surface and fixed with a cyanoacrylic adhesive (23). Clinical attachment level will be calculated as REC + PD.

C) Digital measurements All patients will be scanned and their models will be digitalized with an optical 3D measurement system (3Shape, Erlangen, Germany) creating surface tessellation language (STL) files while a bilateral retractor is placed in the mouth and teeth are held lightly in occlusion. The acquired data will be transferred into a digital imaging software (3Shape Trios®, Erlangen, Germany) in which patient name will be substituted for a random ID number in order to anonymize the data. Baseline and corresponding follow-up scans of each clinical case will be then virtually superimposed and matched into one common coordinate system (Geomagic, 3D Systems, Research Triangle Park, NC, USA) using the tool Control X. By using the buccal surfaces of the concerned teeth as reference points for the superpositioning of the different time points (pre-operative and post-operative), this approach will allow for precise evaluation of dimensional soft tissue alterations over time by a blinded examiner. Vestibular depth will be measured from the GM to the point of greatest concavity of the mucobuccal fold.

The digital linear and volumetric measurements and assessment will be performed by a single, calibrated examiner for the surgical. The examiner will be trained on 15 casts with gingival recessions who will not be included in this study. This examination will be repeated 24 h later; differences of ≤0.5 mm in at least 90% of the cases will be considered to be acceptable.

The following measurements will be taken:

All clinical measurements and volumetric evaluations of the soft will be performed at baseline, 3 months and at 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years.
* Periodontally and systemically healthy.
* Presence of Miller class I and II GR defects or class III with no interproximal clinical attachment loss.
* Recession >2mm in depth at the buccal aspect.
* Full-mouth plaque and bleeding score ≤20%.
* No previous periodontal surgery.
* Presence of identifiable CEJ (a step ≤1mm at the CEJ and/or presence of root abrasion, but with identifiable CEJ, will be accepted).

Exclusion Criteria:

* Tobacco smoking of ≥10 cigarettes a day.
* Contraindications for periodontal surgery.
* Medications known to affect the gingiva or interfere with wound healing.
* Pregnancy.
* Active orthodontic therapy.
* caries or restorations in the area to be treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Complete Root Coverage | 6 months
  By using the buccal surfaces of the concerned teeth as reference points for the superimposition of the different time points (pre-operative and post-operative), this approach will allow for the precise evaluation of dimensional soft tissue alterations over time.

SECONDARY OUTCOMES:
Mean Root Coverage | 6 months
  By using the buccal surfaces of the concerned teeth as reference points for the superimposition of the different time points (pre-operative and post-operative), this approach will allow for the precise evaluation of dimensional soft tissue alterations over time.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Nart, DDS PhD, Study Chair — Universitat Internacional de Catalunya
Locations (1):
- International University of Catalunya, Barcelona, Spain